CLINICAL TRIAL: NCT00658190
Title: Internet-Based Cervical Cytology Screening Program
Acronym: IBCCSP
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, David C. Wilbur, MD, Pathologist, Massachusetts General Hospital
Other Study IDs: 2003P-001658; PRO33199 W81XWH-04-C-0083
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2012-04

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer, automation, Internet, telecytology
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women obtaining routine Pap tests for cervical cancer screening

SUMMARY:
The purpose of this study is to assess whether a system that couples automated screening of Pap Tests with transmission of machine selected digital images, and review by cytologists at a remote location, performs to a clinically effective standard of accuracy.

DETAILED DESCRIPTION:
This clinical study uses the automated screening capabilities of the FocalPoint Primary Screening System (BD) for gynecologic cytology specimens (Pap tests) to allow for automated field of view (FOV) selection, digital image capture, and subsequent Internet-based transmission to a custom designed computer-based image reading station. The system utilizes liquid-based cytology preparations (ThinPrep, SurePath). In such a system, no skilled cytology human resources are necessary at the scanning site, and all expertise can be centralized. Pilot studies showed that the task was feasible to a clinically relevant standard of care. Phase 1 trials on preselected and seeded specimens confirmed this clinical standard. The phase 2 trials extend the concept to a prospectively enrolled population of patients from 2 sites (Walter Reed, Mass General) thereby testing the concept in a population of normal disease prevalence. The final phase 3 will be a larger study with intended use design, siting a screening device at the 121st Army Hospital in Korea and interpreting the specimen images in the US. In addition to the reading of the specimens, the system is designed to give immediate "loop closing" results back to each specimen's originating point immediate upon completion of the test.

ELIGIBILITY:
Inclusion Criteria:

* Female presenting to clinic for a Pap test for any reason

Exclusion Criteria:

* Pregnant
* Prisoners
* Mentally unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females presenting to clinics at MGH or WRAMC for a Pap test
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2003-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Cervical cytology abnormal cases | At enrollment
  Identification of abnormalities compared to the initial interpretation

CONTACTS AND LOCATIONS:
Overall Officials: David C. Wilbur, MD, Principal Investigator — MGH; Barabara A Crothers, D.O, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Eichhorn JH, Brauns TA, Gelfand JA, Crothers BA, Wilbur DC. A novel automated screening and interpretation process for cervical cytology using the internet transmission of low-resolution images: a feasibility study. Cancer. 2005 Aug 25;105(4):199-206. doi: 10.1002/cncr.21098. PMID 15937917